CLINICAL TRIAL: NCT02697851
Title: The Effect of Atazanavir/Cobicistat on the Pharmacokinetics of an Oral Contraceptive Containing Ethinylestradiol and Levonorgestrel (Microgynon 30®) in Healthy Women
Brief Title: Pharmacokinetic Effect of Evotaz/Microgynon Co-administration
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient enrolment and "business reasons"
Sponsor: St Stephens Aids Trust (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: SSAT069
Record Dates: First submitted 2016-02-02; First posted 2016-03-03 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: HIV
MeSH Terms: interventions — Ethinyl Estradiol; Levonorgestrel; Atazanavir Sulfate; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Microgynon 30® for 21 days, Followed by Microgynon 30® for 21 days plus Evotaz® for 14 days, Followed by Evotaz® for 14 days
  Interventions: Drug: Microgynon 30®; Drug: Evotaz®
- Group 2 (Experimental): Evotaz® for 14 days followed by 7 days wash-out, Followed by Microgynon 30® for 21 days plus Evotaz® for 14 days, Followed by Microgynon 30® for 14 days (participants may chose to complete a 21 day pack). The total duration of the study is 57 days (+screening and follow up visits) and patients will have 3 intensive pharmacokinetic days on days 14, 35 and 56
  Interventions: Drug: Microgynon 30®; Drug: Evotaz®

INTERVENTIONS:
Drug: Microgynon 30®
  Other Names: Ethinylestradiol/levonorgestrel
Drug: Evotaz®
  Other Names: Atazanavir /cobicistat

SUMMARY:
This study will investigate the pharmacokinetic of evotaz (atazanavir/cobicistat) and microgynon (ethinylestradiol/levonorgestrel ) when administered alone and together. There will be two study arms, who will take the medications in different orders:

GROUP 1: Microgynon 30® for 21 days, Followed by Microgynon 30® for 21 days plus Evotaz® for 14 days, Followed by Evotaz® for 14 days GROUP 2: Evotaz® for 14 days followed by 7 days wash-out, Followed by Microgynon 30® for 21 days plus Evotaz® for 14 days, Followed by Microgynon 30® for 14 days (participants may chose to complete a 21 day pack). The total duration of the study is 57 days (+screening and follow up visits) and patients will have 3 intensive pharmacokinetic days on days 14, 35 and 56.

DETAILED DESCRIPTION:
Protocol Number: SSAT069

EudraCT Number: 2015-004799-30

Name of Investigational Product: Microgynon 30®; Evotaz®

Name of active ingredients: Ethinylestradiol, levonorgestrel; atazanavir, cobicistat

Study title: The effect of atazanavir/cobicistat on the pharmacokinetics of an oral contraceptive containing ethinylestradiol and levonorgestrel (Microgynon 30®) in healthy women

Phase of study: Phase I

Objectives: The objectives of this study are:

Primary

-To assess the pharmacokinetics of ethinylestradiol/levonorgestrel and atazanavir/cobicistat during co-administration in HIV negative female healthy volunteers

Secondary

* To assess the safety and tolerability of ethinylestradiol/levonorgestrel and atazanavir/cobicistat when co-administered to HIV negative female healthy volunteers
* To investigate the association between genetic polymorphisms in drug disposition genes and drug exposure

Study design: 57 days (excluding screening and follow up), open label, cross-over, pharmacokinetic study

Indication: Not applicable

Methodology: Measurements of steady state pharmacokinetic profiles of plasma ethinylestradiol/levonorgestrel and atazanavir/cobicistat

Planned sample size: Up to 30 female healthy volunteers will be enrolled at baseline in order to achieve 18 completing the study

Summary of eligibility criteria: Healthy female participants as determined by medical history, physical examination, 12-lead electrocardiogram, and clinical laboratory evaluations will be eligible to participate in the study. Women of childbearing potential must not be nursing or pregnant. Women of childbearing potential must have a negative pregnancy test at screening.

Number of study centres: One

Duration of treatment: 57 days (excluding screening and follow up visits)

Dose and route of administration: All participants will be administered Microgynon 30® (ethinylestradiol/levonorgestrel 30 micrograms/150 micrograms) and Evotaz® (atazanavir 300 mg/cobicistat 150 mg) as follows:

GROUP 1:

Microgynon 30® for 21 days Followed by Microgynon 30® for 21 days plus Evotaz® for 14 days Followed by Evotaz® for 14 days

GROUP 2:

Evotaz® for 14 days followed by 7 days wash-out Followed by Microgynon 30® for 21 days plus Evotaz® for 14 days Followed by Microgynon 30® for 14 days (participants may chose to complete a 21 day pack)

Criteria for evaluation: Pharmacokinetic parameters of ethinylestradiol/levonorgestrel and atazanavir/cobicistat will be evaluated on blood drawn on day 14, 35 and 56 at 0 (pre-dose), 1, 2, 4, 6, 8, 10, 12, 24 hours post dose

Safety and tolerability of medications will also be assessed by questions, physical examination and laboratory parameters. These will be performed at regular intervals during the drug study.

Primary Endpoint: Steady state plasma concentrations of ethinylestradiol/levonorgestrel and atazanavir/cobicistat during co-administration in HIV negative female healthy volunteers

Secondary End point: Safety and tolerability of the studied drugs during co-administration

Relationship between genetic polymorphisms and exposure to the studied drugs

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following inclusion criteria within 28 days prior to the baseline visit:

  1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements
  2. Non-pregnant, non-lactating females.
  3. Between 18 to 35 years, inclusive
  4. Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive
  5. ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.
  6. Women of childbearing potential (WOCBP) must be using an additional adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 4 weeks after the study (these include only the ones listed below, as no other hormone-based contraception is allowed during the study)

     A female may be eligible to enter and participate in the study if she:
     1. is of non-child-bearing potential defined as physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
     2. is of child-bearing potential with a reliable negative pregnancy test at both Screening and Day 1 with no risk in between and agrees to use one of the following methods of contraception to avoid pregnancy from screening, throughout the study, and for at least 4 weeks after discontinuation of all study medications:

        * Complete abstinence from penile-vaginal intercourse
        * Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide);
        * Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (please note that not all IUDs meet this criterion)
        * Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject;
        * Any other method with published data showing that the expected failure rate is <1% per year and not containing hormones.

     Any contraception method must be used consistently, in accordance with the approved product label and for at least four weeks after discontinuation of IMP.
  7. Willing to consent to their personal details being entered onto the TOPS database
  8. Willing to provide proof of identity by photographic ID at screen and any subsequent visit
  9. Registered with a GP in the UK

Exclusion Criteria:

* Participants who meet any of the following exclusion criteria are not to be enrolled in this study.

  1. Any clinically significant acute or chronic medical illness
  2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
  3. Positive blood screen for hepatitis B surface antigen or C antibody
  4. Positive blood screen for HIV-1 or 2 by antibody/antigen assay
  5. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
  6. Any medical contra-indication to the use of combined oral contraceptives.
  7. History or presence of allergy to oral contraceptives, atazanavir and cobicistat or excipients (sodium methyl parahydroxybenzoate, lactulose, Hypromellose Colloidal silicon dioxide, Silicified microcrystalline cellulose Crospovidone, Magnesium stearate, Polyvinyl alcohol- partially hydrolysed, Macrogol 3350,Titanium dioxide, Talc, Iron oxide red, Iron oxide black, Lactose monohydrate, Magnesium stearate, Gelatine Yellow iron oxide, Indigocarmin (E132), White ink, Shellac,Titanium dioxide (E171), Ammonium hydroxide, Propylene glycol , Simethicone, Hypromellose, Polyvinyl alcohol- partially hydrolysed, Macrogol 3350)
  8. Current or recent (within three months) gastrointestinal disease
  9. Known intolerance of lactose monohydrate, sunset yellow aluminium lake (E110), and patients with galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption
  10. Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study
  11. Exposure to any investigational drug (or placebo) or participation in a clinical study involving the donation of blood samples within three months of first dose of study drug
  12. Use of any medical products containing estrogens and/or progesteron, including IUS, implants etc. for 4 weeks before screening
  13. Use of any other drugs (unless approved by the Investigator), including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug, unless approved/prescribed by the Principal Investigator as known not to interact with study drugs
  14. Females of childbearing potential without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least four weeks after the end of the treatment period

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-07; Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
assess the pharmacokinetics of ethinylestradiol/levonorgestrel and atazanavir/cobicistat during co-administration in HIV negative female healthy volunteers, as measured by Cthrough | 26 to 36 weeks
  Trough concentration (Ctrough) is defined as the concentration at 24 hours after the observed drug dose
assess the pharmacokinetics of ethinylestradiol/levonorgestrel and atazanavir/cobicistat during co-administration in HIV negative female healthy volunteers, as measured by Cmax | 26 to 36 weeks
  Cmax defined as the maximum observed plasma concentration.
assess the pharmacokinetics of ethinylestradiol/levonorgestrel and atazanavir/cobicistat during co-administration in HIV negative female healthy volunteers, as measured by t1/2 | 26 to 36 weeks
  t1/2 = Elimination half-life
assess the pharmacokinetics of ethinylestradiol/levonorgestrel and atazanavir/cobicistat during co-administration in HIV negative female healthy volunteers, as measured by Tmax | 26 to 36 weeks
  Tmax = time point at Cmax
assess the pharmacokinetics of ethinylestradiol/levonorgestrel and atazanavir/cobicistat during co-administration in HIV negative female healthy volunteers, as measured by total drug exposure | 26 to 36 weeks
  Total drug exposure is expressed as the area under the plasma concentration-time curve from 0-24 hours after dosing (AUC0-24h)

SECONDARY OUTCOMES:
assess the safety and tolerability of the studied drug when co-administered to HIV negative female healthy volunteers, assessed by Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events | 26 to 36 weeks
  studied drug: ethinylestradiol/levonorgestrel and atazanavir/cobicistat
investigate the association between genetic polymorphisms in drug disposition genes and drug exposure as measured by Peak plasma concentration (Cmax) | 26 to 36 weeks
  investigate the association between genetic polymorphisms in drug disposition genes and drug exposure
investigate the association between genetic polymorphisms in drug disposition genes and drug exposure as measured by trough concentration (Ctrough) | 26 to 36 weeks
  investigate the association between genetic polymorphisms in drug disposition genes and drug exposure
investigate the association between genetic polymorphisms in drug disposition genes and drug exposure as measured by Area under the plasma concentration versus time curve (AUC) | 26 to 36 weeks
  investigate the association between genetic polymorphisms in drug disposition genes and drug exposure

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's Centre, Chelsea and Westminster Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided